CLINICAL TRIAL: NCT03218293
Title: The Recovery of Nerve Function Deficient of Combined Intravenous Thrombolysis and Remote Ischemic Post-conditioning in Acute Ischemic Stroke.
Brief Title: Thrombolysis and RIPC in Acute Ischemic Stroke
Acronym: tripcais
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2016-013
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Acute Ischemic Stroke, Cerebral Embolism and Thrombosis
MeSH Terms: conditions — Ischemic Stroke; Intracranial Embolism; Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): Remote ischemic postconditioning（RIPC）：Patients in the RIPC group not only receive foundational treatment but also have five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm using a RIPC device (IPC-906X; Beijing Renqiao Institute of Neuroscience, Beijing, China) after thrombolysis while in-hospital.
  Interventions: Device: RIPC device (IPC-906X)
- Blank control group(BC) (No Intervention): Blank control group:Patients in the BC group only receive foundational treatment, including free radical elimination in the acute stage, blood pressure and blood glucose stabilization, and antiplatelet (aspirin, 100-300 mg/d) and lipid-lowering (atorvastatin, 20 mg/d) drugs,throughout the 14 days in-hospital period without remote ischemic postconditioning after thrombolysis.

INTERVENTIONS:
Device: RIPC device (IPC-906X) — Patients in the RIPC group had five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm after thrombolysis.
  Other Names: Thrombolysis
  Arms: RIPC

SUMMARY:
Remote ischemic postconditioning (RIPC) is suggested to protect the cerebral cell against ischemia in various settings. However, the effect of RIPC in patients with acute ischemic stroke who undergo thrombolysis has yet to be examined. In this single-center, randomized controlled trial, we examined the effect of RIPC on the resolution of nerve function deficient in response to thrombolysis. Patients in the RIPC group had five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm after thrombolysis. The primary endpoint was the recovery of nerve function deficient assessed by National Institutes of Health Stroke Scale(NIHSS), Activities of Daily Living(ADL), Modified Rankin Scale(mRS), CT cerebral perfusion imaging (CTP) and CT angiography(CTA). Secondary endpoints included the following: angiogenesis assessed by the level of vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF).

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Guideline of Thrombolysis in Acute Ischemic Stroke and accomplish intravenous thrombolytic therapy using alteplase;
* The consciousness of patients are conscious,somnolence,confusion and stupor，can comply better with the RIPC treatment;
* Acute ischemic stroke confirmed by cranial CT/MRI;
* Provision of written informed consent.

Exclusion criteria:

* History of cerebral embolism,cerebral hemorrhage, brain tumor, brain trauma or other brain lesion;
* Severe cardiac, liver, or kidney disease, malignancy, systemic organ dysfunction;
* Blood pressure <90/60 mmHg or >200/110 mmHg after treatment;
* Dementia or mental illness;
* History of major surgery or trauma 4 weeks prior to admission;
* Failure to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
the percentage of patients with a favorable outcome, defined as a score of 0 or 1 on the modified Rankin scale (mRS). | Day 90

SECONDARY OUTCOMES:
the percentage of functional recovery at discharge and at day 90, as measured by the NIHSS, the Barthel index (BI) and the mRS | Day 90 and at discharge(up to day 14)
  we measured how many patients achieved a score of 0 or 1 for the NIHSS, 95 for the BI, and 0 - 2 for the mRS.
Plasma biomarker concentrations | Day 1 and at discharge ( up to day 14)
  Venous blood was drawn before the administration of IV tPA and at the end of hospitalization to determine the effect of repeated RIPC on anti-inflammatory (S100-β), vascular (VEGF, bFGF), anti-edema (MMP9), anti-oxidants (OH1) and other pathways (BDNF, HSP).

OTHER OUTCOMES:
mortality rate | up to 3 months.
  three-month mortality rate
the rate of symptomatic hemorrhagic transformation | up to 36 hours
  Defined by European Cooperative Acute Stroke Study III classification
Early neurological deterioration | up to 24 hours after IV tPA
The tolerance index | up to 14 days
  the proportion of patients that could complete every RIPC treatment session during his/her hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Guogang Luo, MD, PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] An JQ, Cheng YW, Guo YC, Wei M, Gong MJ, Tang YL, Yuan XY, Song WF, Mu CY, Zhang AF, Saguner AM, Li GL, Luo GG. Safety and efficacy of remote ischemic postconditioning after thrombolysis in patients with stroke. Neurology. 2020 Dec 15;95(24):e3355-e3363. doi: 10.1212/WNL.0000000000010884. Epub 2020 Oct 7. PMID 33028663